CLINICAL TRIAL: NCT00658411
Title: A Pilot Study of Deferoxamine Before and During Myeloablative Allogeneic Stem Cell Transplantation for Patients With Myelodysplastic Syndromes or Acute Leukemia and Iron Overload
Brief Title: Deferoxamine for Iron Overload Before Allogeneic Stem Cell Transplantation
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Closed due to slow patient accrual
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Philippe Armand, MD, PhD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 07-411
Record Dates: First submitted 2008-03-31; First posted 2008-04-15 (Estimated); Results first posted 2013-04-09 (Estimated); Last update posted 2013-04-09 (Estimated); Status verified 2013-04

CONDITIONS: Acute Myeloid Leukemia; Acute Lymphoblastic Leukemia; Myelodysplastic Syndrome
Keywords: AML; ALL; MDS; iron overload; deferoxamine
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Myelodysplastic Syndromes; Iron Overload | interventions — Deferoxamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- All patients (Experimental): Deferoxamine for >=2 weeks prior to stem cells
  Interventions: Drug: deferoxamine

INTERVENTIONS:
Drug: deferoxamine — Given intravenously or subcutaneously over 8-12 hours daily for at least three weeks prior to transplantation date and continue until the day before the participant receives their donor's stem cells.
  Other Names: Desferal; deferoxamine mesylate

SUMMARY:
The objective of this research study is to determine the safety and feasibility of chelation therapy with deferoxamine for patients with iron overload who are receiving a stem cell transplant. Patients who have iron overload prior to stem cell transplantation may have more toxicity from the transplantation procedure, and thus may benefit from an attempt at iron chelation pre- and peri-transplantation. In this study we are examining the use of deferoxamine starting 2 weeks to 3 months prior to transplantation and continuing through the preparative regimen.

DETAILED DESCRIPTION:
See above

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Histologically confirmed acute myeloid leukemia, acute lymphoblastic leukemia, or myelodysplastic syndrome
* Planned allogeneic stem cell transplantation with myeloablative conditioning regimen; the planned date of transplantation must be at least 4 weeks from time of enrollment
* Severe iron overload as defined by BOTH: Ferritin greater than 1000ng/ml (at the time of donor availability) and Liver iron content estimated greater than or equal to 5mg/g dry weight by MRI (at the time of donor availability)
* Patients with a history of prior autologous transplantation will be eligible for this study

Exclusion Criteria:

* Contraindication to magnetic resonance imaging (MRI)
* Creatinine >2.0mg/dl or creatinine clearance <50ml/min
* Active uncontrolled bacterial or fungal infection
* History of mucormycosis
* Pre-existing clinically apparent retinal neuropathy. If patients have clinically apparent visual loss at the time of screening, they will be excluded if either they have known retinal neuropathy or if this cannot be excluded by further testing
* Pre-existing clinically apparent sensorineural hearing loss. If patients have auditory loss at the time of screening, they will be excluded if either they have known sensorineural hearing loss, or if this cannot be excluded by further testing
* Pregnancy or inability or unwillingness to use contraception during the time of the study
* Lactating patients
* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2008-08; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Armand, MD, PhD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

REFERENCES:
- [Derived] Armand P, Sainvil MM, Kim HT, Rhodes J, Cutler C, Ho VT, Koreth J, Alyea EP, Neufeld EJ, Kwong RY, Soiffer RJ, Antin JH. Pre-transplantation iron chelation in patients with MDS or acute leukemia and iron overload undergoing myeloablative allo-SCT. Bone Marrow Transplant. 2013 Jan;48(1):146-7. doi: 10.1038/bmt.2012.94. Epub 2012 May 21. No abstract available. PMID 22609885

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult patients with AML, ALL, MDS scheduled for HSCT with myeloablative conditioning, who in addition were found to have both a serum ferritin ≥ 1000 ng/ml and a liver iron content (LIC) > 5 mg/g dry weight (mg/gdw) based on hepatic T2* measurement, were offered enrollment on the chelation study.
Groups:
- All Patients: Deferoxamine for >= 2 weeks prior to stem cells
Period: Overall Study
Arm/Group | All Patients
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- All Patients: Deferoxamine prior to stem cells
Arm/Group | All Patients
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 48 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Safety of Deferoxamine Therapy Determined by the Number of Participants With Grade 3 or Higher Toxicities.
Description: All patients meeting the criteria for Severe iron overload as defined by BOTH:
  ferritin ≥ 1000 ng/ml and liver iron content(LIC) ≥ 5 mg/gdw were enrolled and received chelation therapy with Deferoxamine. All patients who received chelation therapy were monitored for grade 3 or above toxicity Attributable to Deferoxamine(grades defined by the CTCAE Version 3). The number of participants with grade 3 or higher toxicities were measured and used to determine the safety of chelation therapy.
Time Frame: Baseline , 6 month, 1 year
Population: Patients who met criteria for iron overload pre-transplant, as defined by the protocol, were enrolled on study for chelation therapy. Those patients who received therapy were monitored for toxicities using the CTCAE version 3.0.
Measure: Number; unit: Participants
Groups:
- Deferoxamine: All patients received a maximum dose of 50mg/kg/d of deferoxamine as chelation therapy for at least 2 weeks prior to receiving myeloablative transplant.
Arm/Group | Deferoxamine
Number analyzed (Participants) | 5
Participants
  Baseline | 5 (9.8) [20 to 52]
  6 month | 0
  1 year | 0

2. Secondary Outcome: 1-year Post-Transplant Survival
Description: Survival information for the 5 patients who were treated with deferoxamine was collected. This information was used to determine transplant-related mortality, relapse, disease-free and overall survival.
Time Frame: 1 year
Population: Stopped early for poor accrual
Measure: Number; unit: participants
Groups:
- Transplant-Related Mortality (Deferoxamine): Patients who received Deferoxamine and passed away as a result of transplant or study treatment without prior relapse at 1 year.
- Relapse (Deferoxamine): Patients who received Deferoxamine and relapsed post transplant at 1 year.
- Disease-Free Survival (Deferoxamine): Patients who received Deferoxamine and are currently alive without incidence of relapse at 1 year.
- Overall Survival (Deferoxamine): Patients who received Deferoxamine and have relapsed and is alive at 1 year.
Arm/Group | Transplant-Related Mortality (Deferoxamine) | Relapse (Deferoxamine) | Disease-Free Survival (Deferoxamine) | Overall Survival (Deferoxamine)
Number analyzed (Participants) | 5 | 5 | 5 | 5
participants | 0 | 0 | 5 | 0

ADVERSE EVENTS:
Time Frame: All patients were monitored for toxicities from the time of chelation to study completion (1 year post transplant).
Arm/Group | Deferoxamine
Serious Adverse Events (participants affected / at risk) | 1/5
Other Adverse Events (participants affected / at risk) | 0/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Deferoxamine (N=5)
Hypotension (Vascular disorders) | 1 (5) — Transient hypotension requiring vasopressor support

LIMITATIONS AND CAVEATS:
The number of patients enrolled on this study is far too small to draw reliable conclusions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes